CLINICAL TRIAL: NCT04404725
Title: Comparing Biofinity Toric Multifocal to Ultra Multifocal for Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-110
Record Dates: First submitted 2020-05-22; First posted 2020-05-27 (Actual); Results first posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Astigmatism; Presbyopia
MeSH Terms: conditions — Astigmatism; Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- comfilcon A then samfilcon A (Experimental): Subjects were randomized to wear comfilcon A for one month then Samfilcon A for one month in this randomized, bilateral cross-over study.
  Interventions: Device: comfilcon A; Device: Samfilcon A
- samfilcon A then comfilcon A (Active Comparator): Subjects were randomized to wear samfilcon A for one month then comfilcon A for one month in this randomized, bilateral cross-over study.
  Interventions: Device: comfilcon A; Device: Samfilcon A

INTERVENTIONS:
Device: comfilcon A — Subjects will be randomized to wear comfilcon A for one month.
  Other Names: Biofinity Toric Multifocal
Device: Samfilcon A — Subjects will be randomized to wear samfilcon A for one month.
  Other Names: Ultra Multifocal for Astigmatism

SUMMARY:
The objective of the study was to compare the handling and performance of Biofinity Toric Multifocal to Ultra Multifocal for Astigmatism.

DETAILED DESCRIPTION:
The objective of the study was to compare the handling and performance of Biofinity Toric Multifocal to Ultra Multifocal for Astigmatism. This is a prospective, randomized, participant masked, crossover, bilateral dispensing study.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 42 years of age and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Self reports having a full eye examination in the previous two years;
4. Anticipates being able to wear the study lenses for at least 8 hours a day, 5 days a week;
5. Is willing and able to follow instructions and maintain the appointment schedule;
6. Habitually wears soft contact lens for the past 3 months minimum;
7. Has refractive astigmatism of at least -0.75DC;
8. Is presbyopic and requires a reading addition of at least +0.75D;
9. Can be fit and achieve binocular distance vision of at least 20/30 Snellen (or +0.20 logMAR) which participants also deem to be 'acceptable', with the available study lens parameters (sphere +4 to -6; cylinder -0.75 to -1.75DC; near addition +0.75 to +2.50).

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Habitually wears one of the study contact lenses;
3. Has any known active* ocular disease and/or infection;
4. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
5. Is using any systemic or topical medications that in the opinion of the investigator may affect contact lens wear or a study outcome variable;
6. Has known sensitivity to the diagnostic sodium fluorescein and/or the care product Opti-Free PureMoist being used in the study;
7. Self-reports as pregnant, lactating or planning a pregnancy at the time of enrolment;
8. Has undergone refractive error surgery. * For the purposes of this study, active ocular disease is defined as infection or inflammation which requires therapeutic treatment. Mild (i.e. not considered clinically relevant) lid abnormalities (blepharitis, meibomian gland dysfunction, papillae), corneal and conjunctival staining and dry eye are not considered active ocular disease. Neovascularization and corneal scars are the result of previous hypoxia, infection or inflammation and are therefore not active.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD FCOptom, Principal Investigator — University of Waterloo; Fiona Soong, Principal Investigator — Eyes on Sheppard Clinic; Adam Keech, Principal Investigator — Oakley Eyecare; Howard Dolman, Principal Investigator — Dolman Eyecare Centre; Kristin Heeney, Principal Investigator — Spadina Optometry; Michael Kreuzer, Principal Investigator — Glasses Half Full; Shane Foster, Principal Investigator — Athens Eye Care; Michael Cymbor, Principal Investigator — Nittany Eye Associates
Locations (7):
- United States (2):
  - Athens Eye care, Athens, Ohio
  - Nittany Eye Associates, State College, Pennsylvania
- Canada (5):
  - Glasses Half Full, Edmonton, Alberta
  - Oakley Eyecare, Winnipeg, Manitoba
  - Dolman Eyecare Centre, New Hamburg, Ontario
  - Spadina Optometry, Toronto, Ontario
  - Lyndon Jones, Waterloo, Ontorio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 64 eligible participants, 63 were dispensed with study products, and one participant withdrew after the screening visit due to lens handling and general time commitment concerns.
Period: First Intervention
Arm/Group | Comfilcon A Then Samfilcon A | Samfilcon A Then Comfilcon A
Started | 32 | 31
Completed | 32 | 29
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: Second Intervention
Arm/Group | Comfilcon A Then Samfilcon A | Samfilcon A Then Comfilcon A
Started | 32 | 29
Completed | 31 | 27
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects were randomized to wear comfilcon A for one month then Samfilcon A for one month in this randomized, bilateral cross-over study. The baseline measures include information of all 64 eligible participants.
  Of the 64 eligible participants, 63 were dispensed with study products, and one participant withdrew after the screening visit due to lens handling and general time commitment concerns.
Arm/Group | Overall Study
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 64
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 48
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Ease of Lens Handling at Insertion
Description: Subjective at-home ratings for ease of lens handling for insertion, using a 0-10 scale (0-Very difficult, 10 - Very easy).
Time Frame: Day 28
Population: Out of 58 subjects who completed the study, data of three participants from the comfilcon A Arm /group and data of two participants from samfilcon A Arm / group was excluded from the analysis due to minor protocol deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Comfilcon A: Subjects were randomized to wear comfilcon A for one month in this randomized, bilateral cross-over study.
- Samfilcon A: Subjects were randomized to wear samfilcon A for one month in this randomized, bilateral cross-over study.
Arm/Group | Comfilcon A | Samfilcon A
Number analyzed (Participants) | 55 | 56
score on a scale | 8.6 (1.6) | 8.8 (1.8)

ADVERSE EVENTS:
Time Frame: One month on each study lenses, a total of two months.
Arm/Group | Comfilcon A | Samfilcon A
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/63
Other Adverse Events (participants affected / at risk) | 9/61 | 9/63
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Comfilcon A (N=61) | Samfilcon A (N=63)
conjunctivitis (Eye disorders) | 5 (5) | 5 (5)
Infiltrative Keratitis (Eye disorders) | 2 (2) | 0 (0)
Non-Ocular Event (General disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT04404725/Prot_SAP_000.pdf